CLINICAL TRIAL: NCT05930795
Title: Evaluation of the Comparison of Anatomical and Functional Results of Laparoscopic Pectopexy and Laparoscopic Lateral Suspension Surgeries for the Treatment of Pelvic Organ Prolapse
Brief Title: Comparison of Laparoscopic Pectopexy and Laparoscopic Lateral Suspension Surgeries
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gaziosmanpasa Research and Education Hospital (Other Government)
Responsible Party: Principal Investigator, Serkan Kumbasar, Principal Investigator, Gaziosmanpasa Research and Education Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: GaziosmanpaşaTREHv
Record Dates: First submitted 2023-06-02; First posted 2023-07-05 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Patients With Pelvic Organ Prolapse; Pectopexy; Lateral Suspension; Pop-q; Pisq-12

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients with pelvic organ prolapse undergone pectopexy surgery (Active Comparator)
  Interventions: Procedure: pectopexy
- Patients with pelvic organ prolapse undergone lateral suspension surgery (Active Comparator)
  Interventions: Procedure: lateral suspension

INTERVENTIONS:
Procedure: pectopexy — pectopexy: surgery performed by suspending prolapsed uterus or vault to the pectineal ligament
  Other Names: surgery performed by suspending prolapsed uterus or vault to the pectineal ligament
  Arms: Patients with pelvic organ prolapse undergone pectopexy surgery
Procedure: lateral suspension — lateral suspension: surgery performed by suspending prolapsed uterus or vault to the lateral walls of the abdomen corresponding to the 3 cm anterior superior to the iliac crest
  Arms: Patients with pelvic organ prolapse undergone lateral suspension surgery

SUMMARY:
There is not a study in the literature comparing laparoscopic pectopexy and laparoscopic lateral suspension (LLS) surgeries in the surgical treatment of pelvic organ prolapse. However, there are studies comparing the efficacy of other surgery types for pelvic organ prolapse. For example,In a study, the clinical and anatomical success rate in LLS operations was 83.8%, while the success rate in abdominal sacropexy operation was 89.2%.In another study in which pectopexy and vaginal sacro spinous fixation operations were compared, apical prolapse recurrence rates were found to be similar in both groups.

DETAILED DESCRIPTION:
Pelvic organ prolapse (POP) can be defined as the protrusion of the pelvic organs out of the vagina. Many women experience the symptoms of prolapse of the pelvic organs during their daily activities, during sexual intercourse or during exercise. POP causes various undesirable effects in terms of sexual life and body aesthetics in women. With the increase in the number of elderly individuals in societies, the prevalence of prolapse cases is increasing and is becoming more common.

Patients who had laparoscopic pectopexy operation due to minimum POPQ stage 2 according to the International Classification of Pelvic Organ Prolapse Quantification (POP Q) in our hospital and who had ls lateral suspension surgery with the same indication were planned to be included retrospectively. In the first group, patients who had laparoscopic pectopexy operation were planned to be included. In the second group, it was planned to include patients who had ls lateral suspension operation.

Demographic and intra operative data collected before the procedure: (operation time, estimated blood loss, hospital stay, bowel and bladder injury) and intra operative and postoperative complications and recurrence rates and anatomically preoperative and post op Pelvic prolapse (with POP-Q classification), PopQ values (minimum 6 months) were aimed to be compared between two groups to assess anatomic comparement. Furthermore, the patients will be called back and Pelvic Organ Prolapse / Incontinence Sexual Questionnaire (PİS-Q) questionnaire will be applied to both groups and the results will be compared prospectively to assess functional results.

ELIGIBILITY:
Inclusion Criteria:

* Patients with POP Q stage 2 and above, operated for symptomatic pelvic organ prolapse,

  * Being a Citizen of the Republic of Turkey over the age of 18
  * Patients operated by the same experienced surgeons

Exclusion Criteria:

* To have received chemotherapy and/or radiotherapy for any reason before
* Having previously operated for prolapse
* Cases with Contraindications for Laparoscopy
* Cases with severe cardiovascular or respiratory disease

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2022-08-10 (Actual); Primary Completion 2023-08-10 (Actual); Study Completion 2023-09-10 (Actual)

PRIMARY OUTCOMES:
Comparison of pre and post operative assessment of POP-Q measurements | 1 year
  Comparison of POP-Q values of patients undergone pectopexy and lateral suspension pre and postoperatively.
Comparison of Pre and post operative assessment of Pelvic Organ Prolapse / Incontinence Sexual Questionnaire | 1 year
  Units on a scale of the patients obtained with Pelvic Organ Prolapse / Incontinence Sexual Questionnaire will be compared before and after surgery. PISQ- 12 is a Likert type of survey with five options (scoring from 0 to 4) in each question and the patient is asked a total of 12 questions. The total score is calculated by summing points given to each question. A higher score means better sexual function and the highest total score is 48.

CONTACTS AND LOCATIONS:
Locations (1):
- Gaziosmanpasa Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided